CLINICAL TRIAL: NCT05646784
Title: Pathophysiological Aspects of the Role of Inflammation and Gut Microbiota in Mood Disorders, and Their Therapeutic Implications in Lebanese Population
Brief Title: Gut Microbiota in Mood Disorders in Lebanese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Joseph University, Beirut, Lebanon (Other)
Collaborators: Lallemand Health Solutions, Canada (Unknown)
Responsible Party: Principal Investigator, Nassim Fares, Full Professor of Physiology, head of the research lab of physiology & pathophysiology, St Joseph University, Beirut, Lebanon
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: CEHDF2009
Record Dates: First submitted 2022-11-22; First posted 2022-12-12 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Gut Microbiome; Mood Disorders
Keywords: Gut Microbiome; mood disorders; Lebanon; Depression
MeSH Terms: conditions — Mood Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A double-blind randomized probiotic versus placebo clinical trial will be performed on the target population under medical secured environment. A re-evaluation of the gut bacterial profile, inflammatory markers and depression scoring will be performed at the end of the study. Depression score at baseline and at the end using the same scoring test (MADRS) will be assessed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cerebiome for Depressive patient (Experimental): Patients in a current episode of MDD, as determined by the Mini International Neuropsychiatric Interview (MINI) per DSM-V criteria recruited from Hôtel-Dieu de France hospital as well as from clinics in North Lebanon.
  Interventions: Drug: Cerebiome
- Placebo for Control group (Placebo Comparator): Second group of patients in a current episode of MDD, as determined by the Mini International Neuropsychiatric Interview (MINI) per DSM-V criteria recruited from Hôtel-Dieu de France hospital as well as from clinics in North Lebanon.
  Interventions: Drug: Placebo
- Healthy control (No Intervention): Healthy control not suffering from any mental condition according to the Mini International Neuropsychiatric Interview (MINI) per DSM-V criteria.
  Healthy volunteers will be recruited from students at the Saint-Joseph and the Lebanese universities.

INTERVENTIONS:
Drug: Cerebiome — Evaluate the effect of oral intake of a probiotic agent on plasma inflammatory markers, gut bacterial profile and depressive state in a subgroup of target patients versus a subgroup treated with placebo
  Arms: Cerebiome for Depressive patient
Drug: Placebo — Placebo effect: Evaluate the effect of oral intake of a placebo, on clinical and plasma inflammatory markers, in a subgroup treated with placebo, in combination with conventional treatment for 12 weeks
  Arms: Placebo for Control group

SUMMARY:
This study aims to evaluate the pathophysiological aspects of the role of inflammation and gut microbiota in mood disorders, in particular in depression, and their therapeutic implications on a cohort of the Lebanese population. Specific objective: The evaluation of probiotic intake (CEREBIOME®, Lallemand Health Solutions Inc., Mirabel, Canada) on the inflammatory state, gut bacterial profile and the depressive state.

Evaluate the effect of oral intake of a probiotic agent on plasma inflammatory markers, gut bacterial profile and depressive state in a subgroup of target patients versus a subgroup treated with placebo, in combination with conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive disorder: current depressive episode according to MINI (DSM-5) with a MADRS score of ≥ 20
* Males and females between ages 18 and 65
* Able to understand and comply with the requirements of the study
* Provision of written informed consent

Exclusion Criteria:

* Patients under anti-inflammatory drugs
* Patients under immuno-suppressants
* Use of any type of laxative
* Women who are pregnant, breastfeeding, or planning to become pregnant during the trial
* Bipolar, schizophrenia, and addiction disorders
* Any antibiotic therapy in the past 4 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Concentration of plasma inflammatory markers | 12 weeks of the start of the treatment
  Blood samples (serum) will be used for the dosage of of markers like CRP, ILs-1, IL-6, and cortisol

SECONDARY OUTCOMES:
Metagenomic analysis of the gut microbiota | 12 weeks of the start of the treatment
  The diversity of the gut microbiota will be assessed by the 16S rRNA gene sequencing technique using PCR to target and amplify portions of the hypervariable regions (V1-V9) of the bacterial 16S rRNA gene. Amplicons from separate samples are then given molecular barcodes, pooled together, and sequenced. After sequencing, raw data is analyzed with a bioinformatics pipeline and comparison to a 16S reference database. After the reads are assigned to a phylogenetic rank, a taxonomy profile can be generated
Depression score | 12 weeks of the start of the treatment
  Improvement of depression will be assessed using the MADRS tool

CONTACTS AND LOCATIONS:
Overall Officials: Nassim Fares, Ph.D; HDR, Principal Investigator — Saint-Joseph University
Locations (1):
- Saint-Joseph University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Capuco A, Urits I, Hasoon J, Chun R, Gerald B, Wang JK, Ngo AL, Simopoulos T, Kaye AD, Colontonio MM, Parker-Actlis TQ, Fuller MC, Viswanath O. Gut Microbiome Dysbiosis and Depression: a Comprehensive Review. Curr Pain Headache Rep. 2020 Jun 6;24(7):36. doi: 10.1007/s11916-020-00871-x. PMID 32506238
- [Background] DAS B, Nair GB. Homeostasis and dysbiosis of the gut microbiome in health and disease. J Biosci. 2019 Oct;44(5):117. PMID 31719226
- [Background] Kim JK, Lee KE, Lee SA, Jang HM, Kim DH. Interplay Between Human Gut Bacteria Escherichia coli and Lactobacillus mucosae in the Occurrence of Neuropsychiatric Disorders in Mice. Front Immunol. 2020 Feb 25;11:273. doi: 10.3389/fimmu.2020.00273. eCollection 2020. PMID 32158447
- [Background] Lamers F, Milaneschi Y, Smit JH, Schoevers RA, Wittenberg G, Penninx BWJH. Longitudinal Association Between Depression and Inflammatory Markers: Results From the Netherlands Study of Depression and Anxiety. Biol Psychiatry. 2019 May 15;85(10):829-837. doi: 10.1016/j.biopsych.2018.12.020. Epub 2019 Jan 9. PMID 30819515
- [Background] Karle IL. Flexibility in peptide molecules and restraints imposed by hydrogen bonds, the Aib residue, and core inserts. Biopolymers. 1996;40(1):157-80. doi: 10.1002/(sici)1097-0282(1996)40:13.0.co;2-v. PMID 8541446
- [Background] Misera A, Liskiewicz P, Loniewski I, Skonieczna-Zydecka K, Samochowiec J. Effect of Psychobiotics on Psychometric Tests and Inflammatory Markers in Major Depressive Disorder: Meta-Analysis of Randomized Controlled Trials with Meta-Regression. Pharmaceuticals (Basel). 2021 Sep 23;14(10):952. doi: 10.3390/ph14100952. PMID 34681176
- [Background] Sanada K, Nakajima S, Kurokawa S, Barcelo-Soler A, Ikuse D, Hirata A, Yoshizawa A, Tomizawa Y, Salas-Valero M, Noda Y, Mimura M, Iwanami A, Kishimoto T. Gut microbiota and major depressive disorder: A systematic review and meta-analysis. J Affect Disord. 2020 Apr 1;266:1-13. doi: 10.1016/j.jad.2020.01.102. Epub 2020 Jan 23. PMID 32056863
- [Background] Sarkar A, Harty S, Lehto SM, Moeller AH, Dinan TG, Dunbar RIM, Cryan JF, Burnet PWJ. The Microbiome in Psychology and Cognitive Neuroscience. Trends Cogn Sci. 2018 Jul;22(7):611-636. doi: 10.1016/j.tics.2018.04.006. Epub 2018 Jun 12. PMID 29907531
- [Background] Tian P, Chen Y, Zhu H, Wang L, Qian X, Zou R, Zhao J, Zhang H, Qian L, Wang Q, Wang G, Chen W. Bifidobacterium breve CCFM1025 attenuates major depression disorder via regulating gut microbiome and tryptophan metabolism: A randomized clinical trial. Brain Behav Immun. 2022 Feb;100:233-241. doi: 10.1016/j.bbi.2021.11.023. Epub 2021 Dec 4. PMID 34875345
- [Background] Winter G, Hart RA, Charlesworth RPG, Sharpley CF. Gut microbiome and depression: what we know and what we need to know. Rev Neurosci. 2018 Aug 28;29(6):629-643. doi: 10.1515/revneuro-2017-0072. PMID 29397391
- [Background] Zunszain PA, Anacker C, Cattaneo A, Carvalho LA, Pariante CM. Glucocorticoids, cytokines and brain abnormalities in depression. Prog Neuropsychopharmacol Biol Psychiatry. 2011 Apr 29;35(3):722-9. doi: 10.1016/j.pnpbp.2010.04.011. Epub 2010 Apr 18. PMID 20406665